CLINICAL TRIAL: NCT05569408
Title: An Observational Study to Assess the Real-world Effectiveness of EVUSHELD™ (Tixagevimab/Cilgavimab) as Pre-exposure Prophylaxis Against COVID-19 Among EVUSHELD-eligible Populations in the United States Department of Defense Healthcare System
Brief Title: eVusheld Assessment reaL wORld Effectiveness in DoD Health System
Acronym: VALOR DoD
Status: Completed | Type: Observational
Sponsor: AstraZeneca (Industry)
Responsible Party: Sponsor
Other Study IDs: D8850R00016
Record Dates: First submitted 2022-10-04; First posted 2022-10-06 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: COVID-19; SARS-CoV-2; 2019 Novel Coronavirus Disease
Keywords: Evusheld; tixagevimab and cilgavimab; Pre-exposure prophylaxis; COVID-19; SARS-CoV-2; Effectiveness
MeSH Terms: conditions — COVID-19 | interventions — cilgavimab and tixagevimab drug combination

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- EVUSHELD Arm: Individuals given EVUSHELD for prophylaxis
  Interventions: Drug: EVUSHELD
- Concurrent Control Arms: Individuals eligible for Evusheld prophylaxis but did not receive EVUSHELD
  Interventions: Drug: EVUSHELD

INTERVENTIONS:
Drug: EVUSHELD — Tixagevimab (AZD8895) and cilgavimab (AZD1061)
  Other Names: AZD7442

SUMMARY:
An AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population treated in DoD Health system.

DETAILED DESCRIPTION:
This a Phase IV observational, secondary data study to assess the effectiveness of Evusheld in preventing COVID-19 infection and severe outcomes using the electronic medical records from the nationwide integrated health system.

The study is designed as an AstraZeneca-sponsored observational, electronic healthcare record (EHR)-embedded retrospective cohort study to assess the real-world effectiveness of EVUSHELD against SARS-CoV-2 infection, COVID-19-related hospitalization, and other COVID-19 related outcomes in the total EUA-eligible patient population in the DoD health system.

ELIGIBILITY:
Inclusion Criteria:

1. Receipt of Evusheld under the FDA EUA for Evusheld
2. Eligibility for Evusheld use under the EUA. -

Exclusion Criteria:

* None

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All EUA-eligible patient population in the Department of Defence health system.
Sampling Method: Non-Probability Sample
Enrollment: 4724 (Actual)
Dates: Start 2023-08-10 (Actual); Primary Completion 2023-12-22 (Actual); Study Completion 2023-12-22 (Actual)

PRIMARY OUTCOMES:
COVID-19 Hospitalisation | up to 6 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19 hospitalizations up to 6 months following its initial administration
All-cause mortality | up to 6 months
  To compare all-cause mortality up to 6 months following the initial dose of EVUSHELD, among subjects who did and did not receive EVUSHELD as PrEP

SECONDARY OUTCOMES:
Documented SARS-CoV-2 infection | Up to 6 and 12 months
  To assess the effectiveness of EVUSHELD as PrEP against SARS-CoV-2 infection
Medically attended COVID-19 | Up to 6 and 12 months
  To assess the effectiveness of EVUSHELD as PrEP against medically attended COVID-19
COVID-19 hospitalisation | Up 12 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19 hospitalisation at 12 month
COVID-19 Intensive Care Unit (ICU) admisssion | Up 6 and 12 months
  To assess the effectiveness of EVUSHELD as PrEP against ICU admission
COVID-19 related mortality | Up to 6 and 12 months
  To assess the effectiveness of EVUSHELD as PrEP against COVID-19-related mortality

CONTACTS AND LOCATIONS:
Locations (1):
- Research Site, Bethesda, Maryland, United States